CLINICAL TRIAL: NCT03854149
Title: A Prospective, Observational, Multicenter Study on the Safety and Efficacy of Apixaban for the Prevention of Thromboembolism in Adults With Congenital Heart Disease and Atrial Arrhythmias: the PROTECT-AR Study
Brief Title: Apixaban in Adults With Congenital Heart Disease and Atrial Arrhythmias: the PROTECT-AR Study
Acronym: PROTECT_AR
Status: Completed | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Collaborators: Onassis Cardiac Surgery Centre (Other); Attikon Hospital (Other); MITERA Children's Hospital (Unknown)
Responsible Party: Principal Investigator, George Giannakoulas, Assistant Professor - MD, PhD, AHEPA University Hospital
Other Study IDs: PROTECT_AR_trial_01102018_v1.0
Record Dates: First submitted 2019-02-23; First posted 2019-02-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Congenital Heart Disease; Atrial Arrhythmia; Thromboembolism; Anticoagulants Causing Adverse Effects in Therapeutic Use
Keywords: Congenital Heart Disease; Atrial Fibrillation; Thromboembolism; NOAC; Apixaban; Atrial arrhythmias
MeSH Terms: conditions — Heart Defects, Congenital; Thromboembolism; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with CHD & non-valvular atrial arrhythmias: Adults with congenital heart disease and non-valvular atrial arrhythmias (atrial fibrillation, atrial flutter or intra-atrial re-entrant tachycardia)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of apixaban for the prevention of thromboembolism in adult patients with congenital heart disease (CHD) and non-valvular atrial arrhythmias (AA)

DETAILED DESCRIPTION:
Adult patients with congenital heart disease (ACHD) represent a rapidly growing population due to the progress of surgical techniques and optimal medical management. Non-valvular atrial arrhythmias (AA) carries a significant burden for long-term morbidity and potentially mortality in ACHD patients. AA occur three times more frequently in ACHD compared to the general population. When complicating ACHD, AA convey a twofold increase in the risk for stroke, contributing to an up to 100-fold higher prevalence of stroke in the ACHD population compared to age-matched healthy controls. At present, the European Society of Cardiology (ESC) Guidelines suggest oral anticoagulation (OAC) in all adult patients with AA and intracardiac repair, cyanosis, Fontan palliation, or systemic right ventricle. In the remaining ACHD patients with AA, OAC is suggested if CHA2DS2-Vasc (congestive heart failure, hypertension, age ≥75 years, diabetes mellitus, stroke/transient ischemic attack, vascular disease, age 65 to 74 years, sex category) score is ≥1 (Class of recommendation IIa, level of evidence C).

Non-vitamin K oral anticoagulants (NOACs) are increasingly preferred over vitamin-K antagonists (VKAs) in most clinical scenarios due to improved safety (with regard to intracranial and other major bleeding) and efficacy (prevention of embolic stroke or systemic embolism) along with the convenience they offer for patients and physicians (fixed dose, no food and drug interactions, no INR monitoring). On the other hand, scarce data is available on the use of NOAC in ACHD.

In order to address this gap in evidence, we propose a prospective multicenter single arm, observational cohort trial, which will provide data on the efficacy and safety of apixaban used for the prevention of thromboembolism in ACHD patients with AA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years.
2. Presence of congenital heart disease (intracardiac repair, cyanosis, Fontan palliation, or systemic right ventricle or other congenital heart disease).
3. Non-Valvular Atrial Arrhythmia (including at least one electrocardiographically documented episode).
4. Signed written informed consent by the patient for participation in the study and agreement to comply with the medication and the follow-up schedule.

Exclusion Criteria:

1. moderate-to-severe mitral stenosis or mechanical valves
2. patient unwilling or unable to complete follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Congenital Heart Disease and Non-Valvular Atrial Arrhythmias who are routinely treated with apixaban (i.e., new or ongoing users) for stroke prevention at any health-care level in Greece
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Stroke, systemic or pulmonary arterial thromboembolism and intracardiac thrombosis. | up to 58 months
  The composite endpoint of all-cause stroke, systemic and pulmonary embolism and intracardiac thrombosis
Major bleeding | up to 58 months
  Defined as clinically overt bleeding that is associated with:
  * A fall in hemoglobin of 2 g/dL or more
  * A transfusion of ≥2 units of packed red blood cells or whole blood
  * Bleeding in a critical site: intracranial, intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, retroperitoneal
  * Death (fatal bleeding)

SECONDARY OUTCOMES:
Transient ischemic attack | up to 58 months
  Defined as new neurologic symptoms or deficit lasting less than 24 hours with no new infarction on neuroimaging (if available).
Myocardial infarction | up to 58 months
  Defined as the detection of a significant rise/fall of Troponin in association with symptoms of ischemia, ECG changes, proof of ischemia on imaging or intracoronary thrombus at angiography. [Fourth definition of myocardial infarction; European Society of Cardiology (ESC) 2018]
Death from cardiovascular causes | up to 58 months
  Cardiovascular deaths were classified as deaths due to: ischemic stroke, hemorrhagic stroke, systemic or pulmonary embolism, other cardiovascular (i.e., myocardial infarction, sudden death, heart failure) and unobserved deaths.
Τhe composite of major and clinically relevant nonmajor bleeding | up to 58 months
  Clinically relevant nonmajor bleeding bleeding=bleeding that is clinically overt, that satisfies none of the additional criteria required for the event to be adjudicated as a major bleeding event, that led to either hospital admission for bleeding, physician-guided medical or surgical treatment for bleeding, or a change in antithrombotic therapy.
Τhe composite of stroke, systemic or pulmonary arterial thromboembolism and intracardiac thrombosis, transient ischemic attack, myocardial infarction, or cardiovascular death | up to 58 months

OTHER OUTCOMES:
General quality of life | Baseline
  Assessed with questionnaire SF-36
Apixaban persistence | up to 58 months
  The proportion of patients who were on apixaban at enrolment and continued receiving apixaban at the end of the study period.
Apixaban adherence | up to 58 months
  Assessed by reviewing electronic pharmacy prescription data

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Giannakoulas, MD, PhD, Study Chair — AHEPA University Hospital
Locations (4):
- Greece (4):
  - Attikon University Hospital, Athens
  - Mitera Children's Hospital, Athens
  - Onassis Cardiac Surgery Centre, Athens
  - AHEPA University Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kartas A, Doundoulakis I, Ntiloudi D, Koutsakis A, Kosmidis D, Rampidis G, Apostolopoulou S, Frogoudaki A, Tzifa A, Avramidis D, Ntzoyvara O, Liori S, Mousiama T, Mouratoglou SA, Karvounis H, Giannakoulas G. Rationale and design of a prospective, observational, multicentre study on the safety and efficacy of apixaban for the prevention of thromboembolism in adults with congenital heart disease and atrial arrhythmias: the PROTECT-AR study. BMJ Open. 2020 Sep 22;10(9):e038012. doi: 10.1136/bmjopen-2020-038012. PMID 32963069